CLINICAL TRIAL: NCT06785636
Title: A Phase 1b/2a, MultiCenter, Open- Label Study of Pocenbrodib as Monotherapy or in Combination With Abiraterone Acetate, Olaparib, or 177Lu-PSMA-617 in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Open-Label Study of Pocenbrodib Alone and in Combination With Abiraterone Acetate, Olaparib, or 177Lu-PSMA-617
Acronym: P300
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pathos AI, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P-300-02-001
Record Dates: First submitted 2024-12-10; First posted 2025-01-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: mCRPC (Metastatic Castration-resistant Prostate Cancer); Genital Neoplasms, Male; Urogenital Neoplasms; Urogenital Cancers; Prostatic Diseases; Prostatic Neoplasms; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Prostate Cancer
Keywords: mCRPC, metastatic castrate resistant prostate cancer, prostate cancer,; Procenbrodib; castration resistant
MeSH Terms: conditions — Genital Neoplasms, Male; Urogenital Neoplasms; Prostatic Diseases; Prostatic Neoplasms; Male Urogenital Diseases; Neoplasms; Neoplasms by Site | interventions — Abiraterone Acetate; olaparib; Pluvicto

STUDY DESIGN:
Intervention Model Description: Phase 1b/2a open-label dose finding study to assess safety, PK, efficacy, PD in patients with mCRPC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Portion (Experimental): Dose level 1: 50 mg QD (5 days on/2 days off) Dose level 2: 100 mg QD (5 days on/2 days off) Dose level 3: 150 mg QD (5 days on/2 days off) Dose level 4: 200 mg QD (5 days on/2 days off) Dose level 5: 250 mg QD (5 days on/2 days off)
  Interventions: Drug: Pocenbrodib
- Phase 2 portion (Experimental): Phase 2 involves Pocenbrodib monotherapy and in combination with abiraterone acetate, olaprib or 177Lu-PSMA0617
  Interventions: Drug: Pocenbrodib; Drug: Cohort 2A (Pocenbrodib monotherapy), Cohort 2B (Pocenbrodib + abiraterone acetate), Cohort 2C (Pocenbrodib + olaparib), Cohort 2D (Pocenbrodib + 177Lu-PSMA-617

INTERVENTIONS:
Drug: Pocenbrodib — Pocenbrodib is a selective oral inhibitor of CBP/p300 bromodomain interaction with acetylated lysines on histones.
Drug: Cohort 2A (Pocenbrodib monotherapy), Cohort 2B (Pocenbrodib + abiraterone acetate), Cohort 2C (Pocenbrodib + olaparib), Cohort 2D (Pocenbrodib + 177Lu-PSMA-617 — Pocenbrodib alone or in combination
  Arms: Phase 2 portion

SUMMARY:
This is a dose-finding study to assess the safety and preliminary antitumor activity of Pocenbrodib alone or with Abiraterone acetate, Olaparib or 177Lu-PSMA-617 in patients with metastatic castration-resistant prostrate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a Phase 1b/2a multicenter, open-label study to confirm the safety, pharmacokinetics (PK), preliminary antitumor activity, and pharmacodynamics (PD) of pocenbrodib for the treatment of participants with mCRPC who have progressed despite prior therapy and have been treated with at least 1 potent anti-androgen therapy (enzalutamide, apalutamide, abiraterone acetate, or darolutamide).

The Phase 1b portion of the study involves pocenbrodib monotherapy at multiple, sequential five rising doses (50, 100, 150, 200, and 250mg) initially using a QD dosing schedule of 5 days on/2 days off. The first dose level (50 mg) will enroll at least 3 participants (with 3 more added if the first 3 participants yield 1 dose-limiting toxicity). Once safety is confirmed through Data Review Committee (DRC), the next higher pocenbrodib dose level cohort can begin enrollment.

If both acceptable safety and minimal threshold of efficacy (predefined as 30% PSA50 are achieved, the sponsor will proceed to Phase 2a.

Phase 2a will enroll participants in each of 4 cohorts: pocenbrodib monotherapy (2A), and 3 combination therapy cohorts: pocenbrodib + abiraterone acetate (2B), pocenbrodib + olaparib (2C), and pocenbrodib + 177Lu-PSMA-617 (2D). All cohorts may enroll in parallel, but each cohort will be evaluated independently for safety and efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

1. ≥18 years of age
2. Histologic documentation of prostate adenocarcinoma
3. Metastatic disease, documented by imaging. Imaging performed within 56 days prior to Screening is acceptable

Key Exclusion Criteria:

1. Current or prior evidence of any small cell or neuroendocrine histology on the most recent prostate biopsy
2. Any liver metastases confirmed by biopsy or evidence of lesions >1 cm consistent with liver metastases on imaging
3. Intervention with any chemotherapy, investigational agent, or other anticancer drug, including enzalutamide, apalutamide, or darolutamide, 14 days prior to Screening or 5 half-live20.
4. Any other serious underlying medical, psychiatric, psychological, familial, or geographical condition, which in the judgment of the Investigator may interfere with study participation and compliance or place the participant at high risk from treatment-related complicationss from the last dose (whichever is shorter)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with prostate issues
Enrollment: 252 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) and recommended Phase 2 dose (RP2D) | 28-day
  DLT, serious adverse events (SAEs), clinically relevant adverse events (AEs), and clinically relevant safety laboratory values
RECIST v1.1 objective response rate (ORR) | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  Proportion of participants with ORR. The response rate will be reported with an exact 95% CI.
Prostate specific antigen (PSA) | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  PSA decline post-treatment = ≥ 30% PSA50. The PSA will be reported with an exact 95% CI.

SECONDARY OUTCOMES:
Maximum Plasma Concentration Observed (Cmax) | At the end of Cycle 1, 2, 3, and 4 (each cycle is 28 days) or until end of treatment, whichever came first
  Characterize the Cmax of pocenbrodib in men with mCRPC
PSA30 | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  30% decrease from baseline in PSA while on treatment
PSA50 | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  50% decrease from baseline in PSA while on treatment
PSA90 | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  90% decrease from baseline in PSA while on treatment
Progression Free Survival (PFS) | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  Radiographic PFS is defined as the time from the first date of pocenbrodib administration to the date of radiographic disease progression as outlined in PCWG3 guidelines or death from any cause.
Time to Progression (TTP) | From date of enrollment until the date of first documented progression as per PCWG3 criteria, without ongoing clinical benefit or unacceptable toxicity or date of death from any cause, which came first, estimated to be 6 months.
  Time to radiographic PFS is defined as the time from the first date of pocenbrodib administration to the date of radiographic disease progression as outlined in PCWG3 guidelines or death from any cause.
Overall Survival (OS) | From date of first study drug dose until the date of date of death from any cause assessed up to approximately 32 months
  OS is defined as the time from the first date of pocenbrodib administration until death from any cause.
Time of Maximum Plasma Concentration Observed (Tmax) | At the end of Cycle 1, 2, 3, and 4 (each cycle is 28 days) or until end of treatment, whichever came first
  Characterize the Tmax of pocenbrodib in men with mCRPC
Terminal Half-Life (T1/2) | At the end of Cycle 1, 2, 3, and 4 (each cycle is 28 days) or until end of treatment, whichever came first
  Characterize the T 1/2 of pocenbrodib in men with mCRPC

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - MemorialCare Orange Coast Medical Center, Fountain Valley, California
  - University of Colorado Health, Aurora, Colorado
  - Mount Sinai Medical Center, Miami, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Duke University medical center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, P.A, Houston, Texas
  - NEXT Oncology - Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Pathos AI, Inc. will determine once safety and preliminary efficacy is defined.